CLINICAL TRIAL: NCT05103176
Title: Leveraging Behavioral State to Enhance Specificity of Non-invasive Brain Stimulation on Motor Circuits
Brief Title: Brain State-dependent Stimulation to Improve Movement
Acronym: BrainSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael Vesia, PhD, Assistant Professor, Movement Science, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00186637; 1R21NS118055-01A1 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-02 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: fMRI; TMS; brain stimulation; theta burst; posterior parietal cortex; motor control; grasping

STUDY DESIGN:
Intervention Model Description: The investigators will use a randomized block design with up to 65 subjects in up to nine sessions. The first session will screen subjects before enrolling subjects into study. Three sessions will collect functional magnetic resonance imaging (fMRI) scans, neurophysiological measures with TMS, and behavioral measures. After a baseline testing session, subsequent sessions over five days will entail rTMS, followed by two assessments to evaluate the effects of stimulation on brain and behavior. rTMS intervention sessions will consist of: (i) Posterior Parietal Cortex (PPC) stimulation alone, (ii) PPC stimulation paired with a grasp task or (iii) vertex stimulation (as a control condition) paired with a grasp task. Duration of study: Approximately 3-4 weeks (depending upon scheduling)
Who Masked: Participant
Masking Description: Subjects will be randomly assigned to one of the 3 arms of the study. Subjects will be blind to which arm they are in, however, will be aware of what is involved within each of the arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- To PPC, with concurrent task (Experimental): This arm will receive intermittent theta bust stimulation to the PPC site while subjects perform a grasp task
  Interventions: Device: TMS; Behavioral: Object directed grasping
- To PPC, without a concurrent task (Experimental): This arm will receive intermittent theta bust stimulation to the PPC site without a concurrent task
  Interventions: Device: TMS
- To vertex, with concurrent task (Experimental): This arm will receive intermittent theta bust stimulation to the vertex site (control condition) while subjects perform a grasp task
  Interventions: Device: TMS; Behavioral: Object directed grasping

INTERVENTIONS:
Device: TMS — A MagPro X100 magnetic stimulator with a 90mm figure-8 coil (MC-B70, MagVenture Inc.) will be utilized to deliver brain stimulation. All participants will receive five consecutive days of stimulation. The 3-minute session of intermittent Theta Burst Stimulation (iTBS) will consist of 10 bursts of high-frequency stimulation (a 2 s train of 3 biphasic waveform pulses at 50 Hz repeated every 200 ms at 80% AMT) repeated every 10 s for a total of 190 s (600 pulses) to the target area. The target area will be located using BrainSight2 neuronavigation system. The baseline structural scan obtained during the scan 1 will be utilized for this localization process.
  Other Names: MagPro X100 TMS system
Behavioral: Object directed grasping — Subjects will perform a precision grip with the right hand towards either a small or large target object positioned in front of them. The illumination of an LED (green or red) will instruct the subject to plan a precision grip towards either a small or large target object positioned in front of them. After ~1 second, the LED will extinguish and cue subjects to execute the intended object-directed hand action. The presentation of the visual stimuli will be synchronized with the iTBS stimulation, which will occur 800ms before the onset of every "GO" cue in order to modulate cortical activity during both the planning and execution phase of the action.
  Arms: To PPC, with concurrent task; To vertex, with concurrent task

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a powerful tool to non-invasively modulate brain circuits, brain plasticity, and behavior. This proposal will test the hypothesis that controlling behavioral state during focal multi-day rTMS of a brain region involved in grasping movements will enhance the functional specificity of the neuromodulation action among distributed brain regions involved in voluntary motor control and concomitantly improve manual dexterity. Results from this study will be used to optimize rTMS therapy for individuals with neuromotor impairments by controlling behavioral state to improve the efficacy of rTMS treatment.

Healthy volunteers that qualify for this study will have motor skill assessments and basic neuromotor testing (using neurophysiology with TMS and functional Magnetic Resonance Imaging (fMRI) scans). Participants will be asked to come in for up to nine sessions that include 1 screening session, 5 consecutive daily rTMS sessions and 3 assessment sessions with resting-state and task-based fMRI, neurophysiology with TMS, and hand motor tasks over the course of 3-4 weeks.

DETAILED DESCRIPTION:
This study will examine a particular type of rTMS, known as theta burst stimulation (TBS), which has been shown to induce longer lasting effects than other forms of rTMS, making TBS an important tool for therapeutic applications. While TBS provides relatively focal stimulation, effects on the brain occur through interconnected networks in ways that are poorly understood. Moreover, stimulation is highly state-dependent, and the use of rTMS in most therapeutic settings, such as the treatment of motor impairments, leaves behavioral state uncontrolled. Augmenting rTMS therapy by inducing specific behavioral states is an attractive idea for improving therapeutic rTMS, but the relevant knowledge base is sparse. To address this critical gap, this exploratory R21 proposal will examine the effects of TBS and behavioral state on brain and motor behavior. The investigators will test the broad hypothesis that when TBS is applied during a controlled behavior state, motor function will be facilitated, compared to stimulation when behavioral state is uncontrolled. The investigators will focus on the posterior parietal cortex (PPC), and associated parietofrontal circuits, which subserve skilled grasp control, an ability known to be impaired in stroke, traumatic brain injury, and other motor disorders. The investigators will collect functional magnetic resonance imaging (fMRI), neurophysiological measures with TMS, and behavioral measures in all subjects for three different interventions.

In Aim 1, the investigators will show improvement in action performance by manipulating the behavioral state during PPC stimulation.

In Aim 2, the investigators will demonstrate modulation of neurophysiological aftereffects of PPC stimulation on motor output by manipulating behavioral state.

In Aim 3, the investigators will assess the relationship between brain connectivity, plasticity and behavior in response to the behavioral state during brain stimulation.

Impact: Results will provide insights into the effects of rTMS and behavioral state on the brain and behavior. This knowledge will lay a mechanistic foundation for future studies to show how controlling behavioral state during rTMS can improve therapeutic efficacy in neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing age cannot be pregnant or trying to become pregnant
* Ability to tolerate small, enclosed spaces without anxiety
* Ability and willingness to give informed consent to participate
* No history of neurological disorder
* Right handed
* English speaking

Exclusion Criteria:

* Are left-handed
* Are younger than 18 or older than 50 years old
* Women who are pregnant, suspect they are pregnant, or are attempting to become pregnant
* Have metal anywhere in the head, excluding the mouth
* Have a pacemaker, deep brain stimulator, vagus nerve stimulator or any other medically implanted device
* Have cochlear hearing implants
* Are taking GABAergic, NDMA-receptor antagonist, or other drug known to influence neural receptors
* Have any of the below conditions that would put participants at increased risk of having a seizure: a personal or family history of seizure/epilepsy, taking prescription drugs that lower the threshold for seizures, recent history of excessive alcohol consumption, history of alcohol addiction/dependence, recent history of recreational drug use, history of drug addiction/dependence
* Have been diagnosed with any of the following: a stroke, brain hemorrhage, brain tumor, encephalitis, multiple sclerosis, Parkinson's disease or Alzheimer's disease, depression in the past 6 months, attention deficit disorder, schizophrenia, manic depressive (bipolar) disorder, normal pressure hydrocephalus or increased intra-cranial pressure, diabetes requiring insulin treatment, any serious heart disorder or liver disease
* Have had a migraine in the past month
* MRI specific exclusion criteria: Any relevant history of open-heart surgery, artificial heart valve, brain aneurysm surgery, braces or extensive dental work, cataract surgery or lens implant, or artificial limb or joint. History of foreign metallic object in the body such as bullets, BB's, pellets, shrapnel, or metalwork fragments. Claustrophobia, have uncontrollable shaking, or cannot lie still for one hour.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share information about this/these trial(s) via timely registration, updates, and results reporting in ClinicalTrials.gov in accordance with NIH policy. De-identified data will be entered into the in ClinicalTrials.gov in accordance with NIH policy within 1 year of the conclusion of the study.
  In accord with NIH regulations, the investigators will make the data and relevant documentation available to other investigators upon acceptance of the main findings from the study for publication. The investigators will share analysis tools as they are developed. Because the collected data are to remain anonymous, only a subject number will identify all data. To further protect the privacy and confidentiality of the data, data and documentation will be made available only under a data-sharing agreement that provides for restrictions for the transferring of data to others and a commitment that the data will be used for research purposes only and not for a profit-making enterprise.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of the conclusion of the study
Access Criteria: No additional access restrictions will be placed on the de-identified data beyond those that are standard for the NIH.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 enrolled participants were excluded from the study after enrollment but prior toassignment of a participant arm/group. This was due to work/schedule changes ofparticipants, fMRI incidental findings that could affect neurological measures,ineligibility for MRI studies, and participant concerns over access to medicalrecords.
Period: Overall Study
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Started | 19 | 18 | 17
Completed | 17 | 16 | 16
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task | Total
Number analyzed (Participants) | 19 | 18 | 17 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 17 | 54
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 15 | 36
  Male | 10 | 6 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 18 | 17 | 16 | 51
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5
  White | 12 | 9 | 10 | 31
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in the Time to Complete the Nine-hole Peg Test (9-HPT) to Immediate Post-intervention
Description: 9-hole peg test (9-HPT) is a manual dexterity measure in which a participant must place 9 pegs in board with 9 holes, and remove all 9 pegs upon the insertion of all 9 pegs. This is completed with one peg at a time, and only one hand is used. For our study, only the right hand was used. The performance is estimated as the time required to complete the task (seconds). A lower time in seconds is indicative of a better score. For percent change in performance, a higher positive percent is indicative improved performance.
Time Frame: Baseline and immediately post-intervention (session 6, up to Day 15), up to 30 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percentage change in 9HPT time
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percentage change in 9HPT time | 7.37 (4.57) | -0.15 (7.60) | -4.68 (8.13)

2. Primary Outcome: Percentage Change in Amplitude of Motor Evoked Potential (MEP) to Immediate Post-intervention.
Description: Motor cortical excitability is measured by electromyography using MEPs (motor evoked potentials) elicited by TMS (Transcranial magnetic stimulation) to a motor hotspot determined before collection of baseline (baseline occurs before intervention) MEP (motor evoked potential) collection. It was assessed in session 1, 3, 4, 5, 6, and 7, although only session 6 is reported here. An increase in MEPs (motor evoked potentials) is indicative of increased cortical excitability. A positive increase in MEP (motor evoked potential) percent change is indicative of increased cortical excitability.
Time Frame: Baseline and immediately post-intervention (session 6, up to Day 15), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: MEP Percent Increase
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
MEP Percent Increase | 78.9 (73.7) | 31.5 (67.8) | 3.7 (51.1)

3. Primary Outcome: Change From Baseline Functional Connectivity to PPC Stimulation Target Within the Cortical Grasping Network to Immediate Post-intervention.
Description: Resting-state connectivity of low frequency BOLD (blood oxygenation level dependent) fluctuations for a seed at the PPC (posterior parietal cortex). The original analysis was a time-series correlation (Pearson's R) of resting state fMRI data between two regions of interest. The Z-score a Fisher's r-to-z transform. 0 for the Z value means that the pearson's correlation was also 0, positive means positive correlation and negative means it was a negative correlation. Therefore, standard deviations above the mean represented greater connectivity between the regions of interest. There were no clinically relevant thresholds to consider. The two time points being compared were scans from session 2 and session 7.
Time Frame: Baseline (scan acquired during session 2) and immediate post-intervention (scan acquired after intervention during session 7, up to day 20), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject, and another was left out due to improper data as a result of head movement in the scanner.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
Z score | 0.154 (0.474) | 0.110 (0.397) | 0.003 (0.306)

4. Primary Outcome: Change From Baseline Blood Oxygen Level-Dependent (BOLD) Activation, Voxelwise in the Cortical Grasp Network to Immediate Post-intervention.
Description: Parietal-frontal cortical grasping network defined by BOLD change during precision force-tracking task. t-test statistics were acquired for BOLD activation (estimated with univariate GLMs within each individual) from scans pre and post (session 2 and 7) with free surfer software. We ran univariate GLMs for each session for each individual that gave regression coefficients (beta values) for each voxel. We calculated a t-stat for each of those beta-values (each person and session we have a t-stat for our contrast of interest at each voxel). We averaged these across region of interest for each person/session. We ran another paired t-test at the group level to test pre vs post differences. SD shows t-stat variability across people in respective groups. A t-stat of 0 shows no BOLD change, a large positive t-stat shows increase BOLD change (increased connectivity, better outcome), and a large negative t-stat shows decrease BOLD change (decreased connectivity, worse outcome) pre vs post.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: t-test statistic
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
t-test statistic | -0.095 (3.221) | -1.395 (3.176) | -0.391 (2.618)

5. Secondary Outcome: Percentage Change in the Time to Complete the Nine-hole Peg Test (9-HPT) to 1-week Post-intervention
Description: as for outcome 1
Time Frame: Baseline and 1-week post intervention (session 8 or 9, approximately 1 week after session 7, up to day 30), up to 30 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percentage change in 9HPT time
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percentage change in 9HPT time | 3.22 (12.09) | 2.36 (10.95) | 2.95 (10.58)

6. Secondary Outcome: Percentage Change in Amplitude of Motor Evoked Potential (MEP) to 1-week Post-intervention.
Description: Motor cortical excitability is measured by electromyography using MEPs (motor evoked potentials) elicited by TMS (Transcranial magnetic stimulation) to a motor hotspot determined before collection of baseline (baseline occurs before intervention) MEP (motor evoked potential) collection. An increase in MEPs (motor evoked potentials) is indicative of increased cortical excitability. A positive increase in MEP (motor evoked potential) percent change is indicative of increased cortical excitability.
Time Frame: Baseline and 1-week post-intervention (during session 8 or 9, approximately 1 week after session 7, up to day 30), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: MEP Percent Increase
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
MEP Percent Increase | 31.1 (75.2) | 10.3 (55.8) | -11.7 (39.5)

7. Secondary Outcome: Change From Baseline Functional Connectivity to PPC Stimulation Target Within the Cortical Grasping Network to 1-week Post-intervention.
Description: Resting-state connectivity of low frequency BOLD (blood oxygenation level dependent) fluctuations for a seed at the PPC (posterior parietal cortex). The original analysis was a time-series correlation (Pearson's R) of resting state fMRI data between two regions of interest. The Z-score a Fisher's r-to-z transform. 0 for the Z value means that the pearson's correlation was also 0, positive means positive correlation and negative means it was a negative correlation. Therefore, standard deviations above the mean represented greater connectivity between the regions of interest. There were no clinically relevant thresholds to consider.
Time Frame: Baseline (scan acquired during session 2) and 1-week post-intervention (scan during session 8 or 9, approximately 1 week after session 7, up to day 30), up to 60 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
Z score | 0.160 (0.490) | -0.051 (0.431) | 0.091 (0.437)

8. Secondary Outcome: Change From Baseline Blood Oxygen Level-Dependent (BOLD) Activation, Voxelwise in the Cortical Grasp Network to 1-week Post-intervention.
Description: Parietal-frontal cortical grasping network defined by BOLD change during precision force-tracking task. t-test statistics were acquired for BOLD activation (estimated with univariate GLMs within each individual) from scans pre and post (session 2 and 8/9) with free surfer software. We ran univariate GLMs for each session for each individual that gave regression coefficients (beta values) for each voxel. We calculated a t-stat for each of those beta-values (each person and session we have a t-stat for our contrast of interest at each voxel). We averaged these across region of interest for each person/session. We ran another paired t-test at the group level to test pre vs post differences. SD shows t-stat variability across people in respective groups. A t-stat of 0 shows no BOLD change, a large positive t-stat shows increase BOLD change (increased connectivity, better outcome), and a large negative t-stat shows decrease BOLD change (decreased connectivity, worse outcome) pre vs post.
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: t-test statistic
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
t-test statistic | 0.333 (2.739) | -2.100 (2.334) | 0.524 (2.655)

9. Secondary Outcome: Change From Baseline Blood Oxygen Level-Dependent (BOLD) Activation, Voxelwise in Whole Brain to Immediate Post-intervention.
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: t-test statistic
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
t-test statistic | -0.095 (3.221) | -1.395 (3.176) | -0.391 (2.618)

10. Secondary Outcome: Change From Baseline Blood Oxygen Level-Dependent (BOLD) Activation, Voxelwise in Whole Brain to 1-week Post-intervention.
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: t-test statistic
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 15 | 16 | 16
t-test statistic | 0.333 (2.739) | -2.100 (2.334) | 0.524 (2.655)

11. Secondary Outcome: Percentage Change in Accuracy to Precision Force-tracking Task to Immediate Post-intervention
Description: The force tracking task measures one's ability to regulate their grip force. For this task, the participant must adjust their grip of an object to move the cursor in order to correspond with a constantly moving target. The outcome of this measure is the squared distance (error) from the cursor to the target in the precision force-tracking task, estimated as the root mean squared error (RMSE). A lower root mean squared error (RMSE) is indicative of better performance and better ability of a participant to regulate their grip force. A higher percent change in root mean squared error (RMSE) accuracy is indicative of better performance and better ability of a participant to regulate their grip force. It was assessed in session 2, 7, and 8/9, although only session 2 and 7 are reported here.
Time Frame: Baseline(during fMRI during session 2) and immediate post-intervention (during fMRI following stimulation during session 7, up to day 20), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percent Change in RMSE Accuracy
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percent Change in RMSE Accuracy | 16.16 (16.42) | 11.89 (11.85) | 12.41 (16.21)

12. Secondary Outcome: Percentage Change in Accuracy to Precision Force-tracking Task to 1-week Post-intervention
Description: The force tracking task measures one's ability to regulate their grip force. For this task, the participant must adjust their grip of an object to move the cursor in order to correspond with a constantly moving target. The outcome of this measure is the squared distance (error) from the cursor to the target in the precision force-tracking task, estimated as the root mean squared error (RMSE). A lower root mean squared error (RMSE) is indicative of better performance and better ability of a participant to regulate their grip force. A higher percent change in root mean squared error (RMSE) accuracy is indicative of better performance and better ability of a participant to regulate their grip force. It was assessed in session 2, 7, and 8/9, although only session 2 and 8/9 are reported here.
Time Frame: Baseline(during fMRI during session 2) and 1-week post-intervention (during fMRI during session 8 or 9, about a week following last intervention, up to day 30), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percent Change in RMSE Accuracy
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percent Change in RMSE Accuracy | 5.08 (71.67) | 9.91 (32.15) | 27.15 (14.27)

13. Secondary Outcome: Percentage Change in the Mean Choice Reaction Time to Immediate Post-intervention
Description: The cRT (2-choice reaction time control task) is a measurement of visuomotor abilities that are non specific to the reach-to-grasp movement. The outcome for this measure is the mean reaction time for subjects responding in the cRT (2-choice reaction time control task), for correct responses. A lower mean reaction time in seconds is indicative of better visuomotor performance (non specific to the reach-to-grasp movement). A positive percent change in cRT (2-choice reaction time control task) is indicative of better visuomotor performance (non specific to the reach-to-grasp movement).
Time Frame: Baseline and immediately post-intervention (session 6, up to Day 15), up to 30 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percent change in cRT
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percent change in cRT | -1.45 (5.97) | 0.72 (5.08) | -0.43 (3.25)

14. Secondary Outcome: Percentage Change in the Mean Choice Reaction Time to 1-week Post-intervention
Description: as for outcome 13
Time Frame: as for outcome 5
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: Percent change in cRT
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
Percent change in cRT | -1.88 (5.48) | 1.91 (6.09) | -0.14 (8.09)

15. Secondary Outcome: Percentage Change in the Normalized Motor Evoked Potential (MEP) Size to Immediate Post-intervention.
Description: Parietal-motor functional connectivity is measured by electromyography using MEPs (motor evoked potentials) elicited by dual-site TMS (Transcranial magnetic stimulation) to the motor hotspot and a parietal region determined at baseline (baseline occurs before intervention), while subjects perform an object-directed grasp/subjects are at rest. An increase in MEPs (motor evoked potentials) is indicative of increased cortical excitability. A positive increase in MEP (motor evoked potential) percent change, or normalized MEP (motor evoked potential), is indicative of increased cortical excitability. It was assessed in session 1, 3, 4, 5, 6, and 7, although only session 6 is reported here.
Time Frame: Baseline and immediately post-intervention (session 6, up to Day 15), up to 60 minutes
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: MEP Percent Increase
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
MEP Percent Increase | 78.9 (73.7) | 31.5 (67.8) | 3.7 (51.1)

16. Secondary Outcome: Percentage Change in the Normalized Motor Evoked Potential (MEP) Size to 1-week Post-intervention.
Description: Parietal-motor functional connectivity is measured by electromyography using MEPs (motor evoked potentials) elicited by dual-site TMS (Transcranial magnetic stimulation) to the motor hotspot and a parietal region determined at baseline (baseline occurs before intervention), while subjects perform an object-directed grasp/subjects are at rest. An increase in MEPs (motor evoked potentials) is indicative of increased cortical excitability. A positive increase in MEP (motor evoked potential) percent change, or normalized MEP (motor evoked potential), is indicative of increased cortical excitability.
Time Frame: as for outcome 6
Population: One participant was left out of data analysis due to being a pilot subject.
Measure: Mean (Standard Deviation); unit: MEP Percent Increase
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
Number analyzed (Participants) | 16 | 16 | 16
MEP Percent Increase | 31.1 (75.2) | 10.3 (55.8) | -11.7 (39.5)

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Arm/Group | To PPC, With Concurrent Task | To PPC, Without a Concurrent Task | To Vertex, With Concurrent Task
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | To PPC, With Concurrent Task (N=19) | To PPC, Without a Concurrent Task (N=18) | To Vertex, With Concurrent Task (N=17)
Mood Alteration (Nervous system disorders) | 0 | 0 | 1 — Grade 1 - Mild mood alteration as subject reported being lightheaded and anxious as a result of TMS making the participant's hand twitch.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05103176/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT05103176/ICF_001.pdf